CLINICAL TRIAL: NCT02465697
Title: An fMRI Study of the Enhancement of Emotion Regulation in Borderline Patients
Brief Title: Changes in the Brain as Borderline Patients Learn to Regulate Their Emotions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: GCO 05-1110
Record Dates: First submitted 2015-06-04; First posted 2015-06-08 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Borderline Personality Disorders; Avoidant Personality Disorders
Keywords: Borderline Personality Disorder; Avoidant Personality Disorder; Brain Imaging
MeSH Terms: conditions — Borderline Personality Disorder; Personality Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- BPD Emotion Regulation Training (Experimental): Guided practice in reappraisal
  Interventions: Behavioral: Reappraisal Training
- BPD Control (No Intervention): no training in reappraisal
- APD Emotion Regulation Training (Experimental): Guided practice in reappraisal
  Interventions: Behavioral: Reappraisal Training
- APD Controls (No Intervention): no training in reappraisal
- Healthy Controls Emotion Regulation Training (Experimental): Guided practice in reappraisal
  Interventions: Behavioral: Reappraisal Training
- Healthy Controls (No Intervention): no training in reappraisal

INTERVENTIONS:
Behavioral: Reappraisal Training
  Other Names: Emotion Regulation Training
  Arms: APD Emotion Regulation Training; BPD Emotion Regulation Training; Healthy Controls Emotion Regulation Training

SUMMARY:
Borderline Personality Disorder (BPD), a prevalent psychiatric disorder found in approximately 2% to 6% of the population and 20% of hospitalized psychiatric patients, has proven quite treatment resistant. This study is designed to determine whether patients with BPD can be trained to improve their ability to regulate their emotions and whether this leads to changes in how their brans regulate emotion.

DETAILED DESCRIPTION:
Borderline Personality Disorder (BPD) is a common psychiatric disorder found in approximately 2% to 6% of the population . It is characterized by intense and rapid mood changes, self-destructive behavior, suicidality, and tumultuous relationships. In additional to the emotional costs of the suffering experienced by borderline patients and their loved ones, BPD patients typically function at a level substantially below that of individuals with comparable intellect. The difficulty controlling emotion, so central to the disorder, has proved a particularly difficult to treat. The present study utilizes the latest neuroimaging findings in BPD to generate new ideas for the psychotherapy of the disorder.

This project builds upon our previous neuroimaging work, which has shown that when BPD patients try to control their emotions by employing a method that healthy people frequently use quite effectively -- taking an emotional distance from what is upsetting - BPD patients are not able to quiet down the part of their brain that sends out emotional alarm signals. The objective of the present study is to determine whether giving BPD patients special training in using this healthy distancing strategy can help them to improve their ability to regulate their emotions and return their brain activity to a more normal pattern. The investigators will do this by using fMRI to record brain activity as BPD subjects try to use distancing to reduce their emotional reactions to upsetting pictures before any training, then to have them receive specific training in the distancing strategy. After this training we will again obtain an fMRI scan to determine whether their pattern of brain activation has normalized and whether they have been able to better reduce their negative reactions to the pictures. If this is effective, it will show that such training may help BPD patients better regulate their emotions and would support a program to further develop and incorporate distancing training into the psychotherapy of BPD patients.

A second objective of the present study is to determine whether the tendency of BPD patients to become increasingly sensitized to negative situations when they are re-experienced (as shown by increased activity of the brain's emotional alarm system), will reduce with additional exposure, as it does in patients with phobias, or will continue to increase. Knowing this can help the therapist plan how to most therapeutically approach disturbing life experiences in the psychotherapy of BPD patients.

This project represents an important step in brain imaging research since it applies information learned about brain activity patterns to develop new approaches to psychotherapy. It addresses a serious, prevalent and difficult to treat disorder.

ELIGIBILITY:
Inclusion Criteria:

* BPD subjects 18 to 50 years old
* Meet criteria for DSM-IV Borderline Personality Disorder, including the DSM-IV criteria for affective instability (criterion #6), and not meet criteria for Schizotypal Personality Disorder (SPD) or AvPD.
* Subjects in the AvPD group meet DSM-IV criteria for AvPD and not for BPD or SPD.
* All subjects will be free of psychotropic medications for 2 weeks (6 weeks for fluoxetine).
* Subjects may be enrolled in psychotherapy

Exclusion Criteria:

* BPD and AvPD subjects will not meet DSM-IV criteria for past or present PTSD, bipolar I disorder, schizophrenia, schizoaffective disorder, substance dependence, head trauma, CNS neurological disease, seizure disorder or current major depression.
* Substance abuse disorder in the prior 6 months
* Significant medical illness
* Pregnancy
* Metallic foreign-bodies that contraindicate MRI

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 169 (Actual)
Dates: Start 2011-09; Primary Completion 2017-09-21 (Actual); Study Completion 2017-09-21 (Actual)

PRIMARY OUTCOMES:
Changes in BOLD signal in brain | baseline and 5 days
  BOLD signal changes at 5 days compared to baseline to measure reappraisal success using fMRI to record brain activity.
Changes in BOLD signal in brain | baseline and 2 weeks
  BOLD signal changes at 2 weeks compared to baseline to measure reappraisal success using fMRI to record brain activity.

SECONDARY OUTCOMES:
Perceived Stress Scale | baseline and 5 days
  Change in Perceived Stress Scale at 5 days compared to baseline
Perceived Stress Scale | baseline and 2 weeks
  Change in Perceived Stress Scale at 2 weeks compared to baseline
State Trait Anger Expression Inventory (STAXI) | baseline and 5 days
  Change in STAXI at 5 days compared to baseline
State Trait Anger Expression Inventory (STAXI) | baseline and 2 weeks
  Change in STAXI at 2 weeks compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Harold W Koenigsberg, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States